CLINICAL TRIAL: NCT07044362
Title: Histotripsy Plus Chemotherapy for Advanced Colorectal Liver Metastasis: A Prospective, Single-Armed Trial
Brief Title: Histotripsy Plus Chemotherapy vs Chemotherapy Alone for Advanced Colorectal Liver Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6224
Record Dates: First submitted 2025-06-23; First posted 2025-06-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer; Liver Metastases; Liver Cancer
Keywords: Histotripsy; Liver-confined; Liver colorectal cancer liver metastasis; Liver-confined colorectal cancer liver metastasis; Chemotherapy; Advanced Colorectal; Advanced Colorectal Liver Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This is a single arm, prospective, non-randomized trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Histotripsy + Chemotherapy (Experimental): All enrolled participants will undergo combined treatment with Histotripsy and chemotherapy without interruption in the chemotherapy.
  Interventions: Device: HistoSonics Edison® System; Drug: Chemotherapy

INTERVENTIONS:
Device: HistoSonics Edison® System — Histotripsy is a novel, totally non-invasive, non-ionizing, and non-thermal ablation technique that mechanically disrupts tumors through precisely controlled acoustic cavitation. Histotripsy is administered via HistoSonics Edison® System.
Drug: Chemotherapy — Chemotherapy (standard of care with first line therapy of base of 5-FU with either oxaliplatin or irinotecan).

SUMMARY:
The goal of this clinical trial is to learn if histotripsy plus chemotherapy works to treat unresectable, bilobar liver- confined colorectal cancer liver metastasis (CRLM). The main question this clinical trial aims to answer is:

• Does the management of this condition with uninterrupted palliative chemotherapy and histotripsy demonstrate improved progression-free survival?

Participants will:

* Receive chemotherapy treatment per standard procedure.
* Undergo histotripsy treatment according to current standard procedures at Cleveland Clinic.
* Occasionally receive Computerized Tomography (CT) scan with and without contrast, give biopsy of treated and untreated liver lesions, and participate in a blood draw of up to 3 teaspoons at each in-person visit.
* Participate in genetic testing, as a part of the standard of care for the treatment.

DETAILED DESCRIPTION:
This is a prospective trial testing the benefits of histotripsy plus chemotherapy for participants with colorectal liver metastasis. Histotripsy has been approved by the FDA with De Novo classification for non-invasive destruction of liver tumors. Up to 100 participants with colorectal cancer liver metastasis will be included.

ELIGIBILITY:
Inclusion Criteria:

* Participants with liver-confined colorectal cancer liver metastasis (CRLM) or participants who have low-volume pulmonary disease along with CRLM
* Participants receiving first line therapy with base of 5-FU with either oxaliplatin or irinotecan, or who are within 3 months of beginning chemotherapy, or participants who have completed chemotherapy treatment within 1 month of the histotripsy evaluation
* Participants who have undergone other liver-directed therapy, such as ablation, embolization
* Participants with multiple unresectable metastases that cannot be completely treated with resection and/or ablation
* Participants aged ≥18 years

Exclusion Criteria:

* Participants with resectable disease
* Participants with non-pulmonary extra-hepatic disease including but not limited to bone or peritoneal metastasis.
* Participants who are not able to tolerate general anesthesia
* Participants who have Childs C Cirrhosis
* Other non-skin malignancy within 2 years of study
* WBC count < 3,000 /uL
* Absolute Neutrophil Count < 1,500 /uL
* History of Non-malignant serious concurrent illness that would increase the risk of histotripsy
* Participants with MSI-High
* Participants aged < 18 years
* Pregnant participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiologic tumor viability | 90 days post-treatment
  As assessed by the degree of short-term local tumor control in Colorectal Liver Metastasis(CRLM)

SECONDARY OUTCOMES:
Rate of Tumor Necrosis | 30 days post-treatment
  Biopsy results will be used to assess the degree of tumor necrosis in treated lesions.
Percentage of Viable Tumor in Lesion | 30 days post-treatment
  Biopsy results will be used to assess the percentage of lesions that have viable tumor.
Infiltration of CD4 | 30 days post-treatment
  Biopsy results will be used to assess the infiltration of CD4.
Infiltration of CD8 | Baseline, 30 days post-treatment
  Biopsy results will be used to assess the infiltration of CD8.
Infiltration of B-cells | 30 days post- treatment
  Biopsy results will be used to assess the infiltration of B-cells.
Infiltration of CD45 | 30 days post-treatment
  Biopsy results will be used to assess the infiltration of CD45.
Infiltration of CD68 | 30 days post-treatment
  Biopsy results will be used to assess the infiltration of CD68.
Infiltration of PD-1 | 30 days post-treatment
  Biopsy results will be used to assess the infiltration of PD-1.
Infiltration of PD-L1 | 30 days after treatment
  Biopsy results will be used to assess the infiltration of PD-L1.
Infiltration of CTLA-4 | 30 days post-treatment
  Biopsy results will be used to assess the infiltration of CTLA-4.
Overall Survival | Up to 24 months post-treatment
  Median overall survival will be measured up to 2 years post treatment.
Progression Free Survival (PFS) | Up to 24 months post-treatment
  The rate of progression free survival will be measured up to 2 years post treatment.
30 day Complications | 30 days post-treatment
  The safety profile of the treatment, as measured by the complications at 30 days.
90 day Complications | 90 days post-treatment
  The safety profile of the treatment, as measured by the complications at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Aucejo, MD, Principal Investigator — Cleveland Clinic, Digestive Disease Institute
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no need for sharing IPD for this clinical trial.